CLINICAL TRIAL: NCT04166318
Title: A Randomized Phase II Study of De-Intensified ChemoRadiation for Early-Stage Anal Squamous Cell Carcinoma (DECREASE)
Brief Title: Lower-Dose Chemoradiation in Treating Patients With Early-Stage Anal Cancer, the DECREASE Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2182; NCI-2019-02259 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2182 (Other: ECOG-ACRIN Cancer Research Group); EA2182 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anal Basaloid Carcinoma; Anal Canal Cloacogenic Carcinoma; Anal Canal Squamous Cell Carcinoma; Anal Margin Squamous Cell Carcinoma; Stage I Anal Cancer AJCC v8; Stage IIA Anal Cancer AJCC v8
MeSH Terms: conditions — Anal Canal Carcinoma; Anus Neoplasms | interventions — Biopsy; Specimen Handling; Capecitabine; Fluorodeoxyglucose F18; Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (standard-dose chemoradiation) (Active Comparator): Patients undergo 28 fractions of intensity-modulated radiation therapy (IMRT). Within 24 hours, patients also receive mitomycin IV over 30 minutes or less on day 1 and either fluorouracil IV over 24 hours on days 1-4 and 29-32 or capecitabine PO BID 5 days per week (Monday - Friday) until completion of IMRT in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/MRI or receive FDG and undergo PET/CT during baseline. Patients undergo CT or MRI on the trial. Patients also undergo tissue biopsy during screening and at the discretion of the treating physician. Additionally, patients undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (de-intensified chemoradiation) (Experimental): Patients undergo 20 or 23 fractions of IMRT. Within 24 hours, patients also receive mitomycin IV over 30 minutes or less on day 1 and either fluorouracil IV over 24 hours on days 1-4 or capecitabine PO BID 5 days per week (Monday - Friday) until completion of IMRT in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/MRI or receive FDG and undergo PET/CT during baseline. Patients undergo CT or MRI on the trial. Patients also undergo tissue biopsy during screening and at the discretion of the treating physician. Additionally, patients undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Receive FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Given IV
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well lower-dose chemotherapy plus radiation (chemoradiation) therapy works in comparison to standard-dose chemoradiation in treating patients with early-stage anal cancer. Drugs used in chemotherapy, such as mitomycin, fluorouracil, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving chemotherapy with radiation therapy may kill more tumor cells. This study may help doctors find out if lower-dose chemoradiation is as effective and has fewer side effects than standard-dose chemoradiation, which is the usual approach for treatment of this cancer type.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether de-intensified chemoradiation for early stage squamous cell carcinoma of the anal canal (SCCA) is able to maintain excellent 2-year disease control of 85% or higher while improving anorectal health-related quality of life (HRQL), compared to standard-dose chemoradiation therapy (CRT), as measured by the change in the Fecal Incontinence Quality of Life scale (FIQoL) instrument coping/behavior domain from baseline to 1 year.

SECONDARY OBJECTIVES:

I. To compare changes in patient-reported HRQL (as per Fecal Incontinence Severity Index [FISI], Patient Reported Outcomes Measurement Information System [PROMIS], International Index of Erectile Function [IIEF], Sexual Function-Vaginal Changes Questionnaire [SVQ], and Vaginal Assessment Scale [VAS]/Vulvar Assessment Scale [VuAS] instruments) between the experimental and control arm.

II. To compare patterns of failure (local and regional relapse versus distant; in-field versus out-of-field of radiation), disease control, and overall survival between experimental and control arm.

III. To correlate vaginal dilator use during radiation delivery with sexual function.

IV. To measure changes in serum total testosterone from baseline to up to 12 months after radiation.

V. To validate the utility of imaging features of inguinal and pelvic lymph nodes obtained prior to treatment as a prognostic indicator that can identify patients with early-stage anal squamous cell carcinoma for whom treatment with de-intensified chemoradiation is appropriate.

VI. To determine the incidence of and predictors for cardiovascular toxicity in patients receiving fluorouracil (5-FU) or capecitabine.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (STANDARD-DOSE CHEMORADIATION): Patients undergo 28 fractions of intensity-modulated radiation therapy (IMRT). Within 24 hours, patients also receive mitomycin intravenously (IV) over 30 minutes or less on day 1 and either fluorouracil IV over 24 hours on days 1-4 and 29-32 or capecitabine orally (PO) twice daily (BID) 5 days per week (Monday - Friday) until completion of IMRT in the absence of disease progression or unacceptable toxicity.

ARM B (DE-INTENSIFIED CHEMORADIATION): Patients undergo 20 or 23 fractions of IMRT. Within 24 hours, patients also receive mitomycin IV over 30 minutes or less on day 1 and either fluorouracil IV over 24 hours on days 1-4 or capecitabine PO BID 5 days per week (Monday - Friday) until completion of IMRT in the absence of disease progression or unacceptable toxicity.

All patients receive fludeoxyglucose F-18 (FDG) and undergo positron emission tomography (PET)/magnetic resonance imaging (MRI) or receive FDG and undergo PET/computed tomography (CT) during baseline. Patients undergo CT or MRI on the trial. Patients also undergo tissue biopsy during screening and at the discretion of the treating physician. Additionally, patients undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 6 weeks, every 3 months for years 1-2, every 6 months for year 3, then annually for years 4-5.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0 (PRE-REGISTRATION)
* Patient must be ≥ 18 years of age
* Patients must be English speaking to participate in the trial. (Please note that this requirement is due to the fact that the quality-of-life studies are mandatory and we currently do not have full translated versions of the questionnaires into other languages)
* Patient must have histologically proven T1-2N0M0 invasive anal canal or anal margin squamous cell carcinoma with tumors measuring =< 4 cm. This may include tumors of non-keratinizing histology such as basaloid, transitional cell or cloacogenic histology. Measurable disease is not required
* Patients who are status/post local excision or excisional biopsy procedure are eligible provided there was tumor involvement of the anal canal and/or anal verge prior to the reaction, if the margins were positive, and/or if the stage is T2N0 based on tumor size before the procedure. This means that patients with T1N0M0 anal margin squamous cell carcinoma who underwent surgical excision with negative margins and no involvement of the anal verge and/or anal canal are not eligible
* Tumor size must be documented based on physical examination including digital rectal exam and/or anoscopy/proctoscopy within 4 weeks prior to Step 0 pre-registration
* Patient's human immunodeficiency virus (HIV) status must be known and documented at baseline

  * NOTE: For patients without a history of HIV infection, it is recommended (but not required) that updated HIV testing be performed within one year of study enrollment
* Patients who are HIV-negative will be registered to Arm R. They must not have lymph nodes that are radiographically-concerning for cancer involvement using computed tomography (CT) and fludeoxyglucose F-18 (FDG) - positron emission tomography (PET)/CT-based criteria

  * NOTE: Patients who are HIV-negative and meet the below criteria may proceed directly to Step 1 Randomization
  * Patients will be considered to be lymph node (LN) positive and thereby not eligible in this study if the lymph nodes meet any of the following criteria:

    * Mesorectal, presacral, internal iliac or obturator LN with:

      * Short axis measuring > 5 mm based on CT/magnetic resonance imaging (MRI) OR
      * Morphologic features of irregular border or central necrosis if assessed on MRI and LN measures > 3 mm OR
      * FDG uptake > blood pool (Deauville 3-5) based on FDG-PET/CT or PET/MRI
    * Internal Iliac and obturator LN with:

      * Short-axis measuring > 7 mm based on CT/MRI OR
      * Morphologic features of irregular border or central necrosis based on CT/MRI OR
      * FDG uptake > blood pool (Deauville 3-5) based on FDG-PET/CT or PET/MRI
    * External Iliac and common Iliac:

      * Short-axis measuring > 10 mm based on CT/MRI OR
      * Morphologic features of irregular border or central necrosis based on CT/MRI OR
      * FDG uptake > blood pool (Deauville 3-5) based on FDG-PET/CT or PET/MRI
  * Inguinal LN (superficial and deep) meeting any of the following criteria will be ineligible unless an fine needle aspiration (FNA) is performed and resulting cytology is negative.

    * Morphologic features of irregular border or central necrosis based on CT/MRI
    * FDG uptake > liver (Deauville 4) based on FDG-PET/CT.
    * Patients who are HIV-negative and have inguinal lymph nodes that do not meet the above criteria must undergo fine needle aspiration and have negative histology to be eligible
* Patients who are HIV-positive will be registered to Arm S. They must meet the eligibility criteria below:

  * A CD4 count >= 200
  * Imaging submitted to ECOG-ACRIN for central review for confirmation of no lymph node involvement
  * No history of acquired immunodeficiency syndrome (AIDS)-related complications within past year other than a history of low CD4+ T-cell count (> 200/mm^3) prior to initiation of combination antiretroviral therapy
  * Patient must be healthy on the basis of HIV disease with high likelihood of near normal life span were it not for the anal cancer
  * Patient MUST receive appropriate care and treatment for HIV infection, including antiretroviral medications when clinically indicated, and should be under the care of a physician experienced in HIV management. Patients will be eligible regardless of antiretroviral medication provided the regimen has been stable for at least 4 weeks
* STEP 1 RANDOMIZATION
* Patient must have met the eligibility criteria as outlined Step 0 Pre-registration
* Patient must have Eastern Cooperative Oncology Group (ECOG) - American College of Radiology Imaging Network (ACRIN) performance status of 0-2
* Patient must have no history of prior chemotherapy for this malignancy
* Patients must not have undergone previous radiation to the pelvis such that overlapping radiation fields would be expected
* Patient must not have had prior potentially curative surgery (i.e. abdominal-perineal resection) for carcinoma of the anus. However, patients who undergo local excision or excisional biopsy are eligible provided they meet inclusion criteria
* Patients with T1N0M0 anal margin squamous cell carcinoma must not have undergone surgical excision with negative margins and no involvement of the anal verge and/or anal canal
* Patient must not be receiving any other standard anti-cancer therapy or experimental agent concurrently with the study drugs
* Patient must not have intercurrent illness including, but not limited to, ongoing or active infection or psychiatric/social situations that, in the judgement of the investigator, would limit compliance with study requirements
* Patient must not have had significant cardiovascular disease including myocardial infarction, unstable angina, stroke, transient ischemic attack, symptomatic coronary artery disease, symptomatic congestive heart failure, or uncontrolled cardiac arrhythmia within 6 months of Step 1 randomization
* Patient must not have a history of a different malignancy unless they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk of recurrence

  * Exceptions to this rule are individuals with cervical cancer in situ, non-melanoma skin cancers, and colon polyps
* Patient must not have active inflammatory bowel disease (patients requiring current medical interventions or who are symptomatic)
* Patients must not have an active autoimmune or connective tissue disease that has required systemic treatment in the past two years (i.e., with the use of modifying agents, corticosteroids, or immunosuppressive drugs) Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients who are on anti-coagulation with warfarin within 2 weeks prior to Step 1 randomization and are considering the use of capecitabine, must use an alternative anti-coagulant

  * NOTE: Low molecular weight heparin is permitted provided the patient's prothrombin time (PT)/international normalized ratio (INR) is < 1.5
* Patients who will receive capecitabine and are on Dilantin for a seizure disorder must have Dilantin levels checked weekly
* Hemoglobin > 10 g/dL (within 2 weeks prior to Step 1 Randomization)
* Platelets >= 100,000/mm^3 (within 2 weeks prior to Step 1 Randomization)
* Absolute neutrophil count >= 1500/mm^3 (within 2 weeks prior to Step 1 Randomization)
* Serum creatinine must be < 1.5 X upper limit of normal (ULN), or calculated creatinine clearance must be > 50 ml/min (within 2 weeks prior to Step 1 Randomization)
* Total bilirubin must be < 2 X ULN (within 2 weeks prior to Step 1 Randomization)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 X institutional ULN (within 2 weeks prior to Step 1 Randomization)
* Albumin >= 3.0 g/dL (within 2 weeks prior to Step 1 Randomization)
* Women must not be pregnant or breast-feeding because the study treatment administered may cause harm to an unborn fetus or breastfeeding child. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to Step 1 Randomization to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use accepted and effective method(s) of contraception or to abstain from sexual intercourse for the duration of their participation in the study and for at least 6 months after the completion of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control in the de-intensified chemoradiation therapy (CRT) arm | Up to 2 years
  An event is local-regional failure, distant metastasis and chemoradiation-related death. Will determine if de-intensified chemoradiation achieves 2-year disease control of 85% or higher while improving anorectal health-related quality of life (HRQL), compared to standard-dose CRT, as measured by the change in the Fecal Incontinence Quality of Life scale (FIQoL) instrument coping/behavior domain from baseline to 1 year. The co-primary endpoints of disease control and FIQoL will be formally assessed in a hierarchical manner with disease control being assessed first. Will be estimated for all treatment arms using the Kaplan-Meier method (1958).
Change in FIQoL in the de-intensified CRT arm | Baseline up to 1 year
  Quality of life analyses, will be compared between arms using a two-sample independent t-tests at a significance level of 0.05 and appropriate longitudinal models will be evaluated to assess the trajectory of HRQL endpoints over time and to evaluate those trajectories between treatment arms. Overall score and change from baseline will be summarized using mean and standard deviation at each time point for each arm.

SECONDARY OUTCOMES:
Changes in patient-reported outcomes | Baseline up to 5 years
  Will compare changes as per Fecal Incontinence Severity Index [FISI], Patient Reported Outcomes Measurement Information System [PROMIS], International Index of Erectile Function [IIEF], Sexual Function-Vaginal Changes Questionnaire [SVQ], and Vaginal Assessment Scale [VAS]/Vulvar Assessment Scale [VuAS] instruments between the experimental and control arm. Quality of life analyses, will be compared between arms using a two-sample independent t-tests at a significance level of 0.05 and appropriate longitudinal models will be evaluated to assess the trajectory of HRQL endpoints over time and to evaluate those trajectories between treatment arms. Overall score and change from baseline will be summarized using mean and standard deviation at each time point for each arm.
Patterns of failure (local and regional relapse versus distant; in-field versus out-of-field of radiation) | Up to 5 years
  Will be compared between experimental and control arm. The cumulative incidence method will be used to estimate local-regional and distant failure rates and the failure rates for the experimental treatment will be compared against the control using a failure specific log rank test.
Disease control | Up to 5 years
  Will be compared between experimental and control arm. Will be estimated for all treatment arms using the Kaplan-Meier method (1958).
Effect of vaginal dilator use during radiation delivery on sexual function | Up to 5 years
  Vaginal dilator use during radiation delivery will be correlated with sexual function.
Change in serum total testosterone | Baseline up to 12 months after radiation
Utility of image features of inguinal and pelvic lymph nodes obtained prior to treatment | Baseline
  Will be validated as a prognostic indicator that can identify patients with early-stage anal squamous cell carcinoma for whom treatment with de-intensified CRT is appropriate.
Incidence of and predictors for cardiovascular toxicity in patients receiving fluorouracil or capecitabine | Up to 5 years
  Rates of grade 3+ adverse events (Common Terminology Criteria for Adverse Events [CTCAE], version [v.] 5) will be estimated using a binomial distribution along with their associated 95% confidence intervals and compared using Fisher's exact test between arms.

OTHER OUTCOMES:
Overall survival | Up to 5 years
  Will be compared between experimental and control arm. Will be estimated for all treatment arms using the Kaplan-Meier method (1958).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Dorth, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (659):
- United States (659):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Mercy Cancer Center, Merced, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Health Central, Ocoee, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - LincolnHealth - Miles Campus and Hospital, Damariscotta, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Sands Cancer Center, Canandiaqua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming